CLINICAL TRIAL: NCT05372679
Title: Clinical Evaluation of the Therapeutic Intra-Vascular Ultrasound (TIVUS™) System for Renal Denervation in Patients With Uncontrolled Stage 2 Hypertension
Brief Title: REDUCED 1 - Renal Denervation Using Ultrasonic Catheter EmitteD Energy Study /
Acronym: REDUCED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SoniVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNS05-001
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Uncontrolled Stage 2 Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-randomized, open-label clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Renal denervation (Experimental): Denervating the sympathetic nerves surrounding the renal vasculature using unfocused ultrasound
  Interventions: Device: Renal denervation

INTERVENTIONS:
Device: Renal denervation — The TIVUS system will be used for renal denervation

SUMMARY:
This is a prospective, multicenter, non-randomized, open-label clinical study of the safety and performance of the TIVUS™ System in subjects with uncontrolled stage 2 hypertension in order to assess the safety and effectiveness of the TIVUS™ System when used for renal artery denervation. The study will assess the acute and chronic safety of the procedure as well as the reduction in 24-hour ambulatory mean systolic blood pressure from baseline to 3 months after the procedure.

DETAILED DESCRIPTION:
Nearly half of adults in the United States (108 million, or 45%) have hypertension defined as a systolic blood pressure ≥ 130 mm Hg or a diastolic blood pressure ≥ 80 mm Hg or are taking medication for hypertension. Hypertension is associated with cardiovascular and renal pathologies and leads to death if not treated appropriately. The cardiovascular risk factor doubles with each 20/10 mm Hg elevation in BP values above 115/75 mm Hg.

The current first-line therapy for hypertension involves change in life-style (i.e., diet and exercise) and various medications. However, only about 1 in 4 treated adults (24%) with hypertension have their condition under control. Thus, they are at increased risk for the major side effects of chronically elevated blood pressure, myocardial infarction, stroke, renal disease and heart failure. High blood pressure was a primary or contributing cause of death for more than 494,873 people in the United States in 2018, and was estimated to affect around 1.13 billion people worldwide and resulted in approximately 10 million deaths worldwide, in 2015.

About half of adults (45%) with uncontrolled hypertension have a blood pressure of 140/90 mm Hg or higher, now defined as Stage 2 hypertension. This includes 37 million U.S. adults. About 30 million adults are recommended to take medication. Almost two out of three of this group (19 million) have a blood pressure of 140/90 mm Hg or higher. The other 17 million adults are taking medications but are unable to lower their blood pressure below 140/90 mm Hg and are thus at increased risk for the risks associated with uncontrolled high blood pressure9. High blood pressure costs the United States about $131 billion each year, averaged over 12 years from 2003 to 2014.

In the past decade, several devices were developed in order to target the autonomic nervous system and lower BP in patients with uncontrolled hypertension. These devices aim to provide additional treatment option for patients who do not respond to antihypertensive medication. These devices target other BP regulating mechanisms such as baroreflex activation, deep brain stimulation carotid body ablation, direct vagus nerve stimulation, cardiac neuromodulation, central iliac arteriovenous coupler as well as other devices are currently under research, however, there is no medical device that has been approved so far.

The Therapeutic Intra Vascular UltraSound (TIVUS™) System is designed for renal artery nerve ablation using transluminal ultrasound (US). The TIVUS™ System is a high intensity, non-focused, ultrasound catheter system, which enables remote, localized, controlled, and repeatable thermal modulation of nerves adjacent to arterial vessel wall for performing safe and effective therapeutic artery sympathetic denervation. The ultrasonic energy is transmitted from a catheter positioned within the artery lumen, while avoiding direct contact with the artery wall.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study obtained from the patient, according to local regulations, prior to initiation of any study mandated procedure.
2. Male or female, ≥ 18 years of age and ≤ 80 years of age at the time of screening.
3. Individual has office systolic blood pressure (SBP) ≥ 140 mm Hg but < 180 mm Hg, and a diastolic blood pressure (DBP) ≥ 90 mm Hg but < 110 mm Hg based on an average of 3 office seated blood pressure readings measured by a manual, automated or semi-automated validated BP monitor, on current medications. 4. Documented mean daytime ABPM systolic blood pressure (SBP) ≥ 135 mm Hg but < 180 mm Hg, after a 4 week stabilization period.

5. Patient is either on at least one anti-hypertensive medication at maximal tolerated dose with a medically documented intolerance to one or more medications, or on three medications where one is a diuretic.

6. Patient is willing and expected to maintain their anti-hypertensive medication regimen for at least 3 months.

7. Patient is able and willing to comply with all study procedures.

Exclusion Criteria:

1. Patient has been previously diagnosed with abnormal renal artery anatomy and/or renal anatomy such as single kidney, other renal development anomaly such as ectopic or horseshoe kidney, or polycystic kidney disease precluding renal denervation therapy as detailed in the angiographic exclusion criteria.
2. Pregnant or breastfeeding women or women planning a pregnancy within 12 months of study enrollment.
3. Patient has an estimated glomerular filtration rate (eGFR) of < 40mL/min/1.73m2 CKD-EPI as calculated using the CKD-EPI 2021 equation.
4. Patients with uncontrolled rapid AF.
5. Patient has had a previous renal denervation procedure.
6. Patients with daytime ABPM mean systolic blood pressure (SBP) > 180 mm Hg.
7. Patient has Type 1 diabetes or poorly controlled Type 2 diabetes (HbA1c > 9%).
8. Patients with history of myocardial infarction, unstable angina pectoris, heart failure, cerebrovascular accident, or widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
9. Patient has a planned major surgery or cardiovascular intervention in the next 6 months.
10. Patient who has undergone a major surgery or cardiovascular intervention in the previous 3 months.
11. Patient has frequent intermittent or chronic pain that results in treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment.
12. Patient is taking immunosuppressive therapy for diseases featuring vasculitis.
13. Patient on anticoagulant therapy that cannot be temporarily withheld for study procedure.
14. Contraindication to recommended denervation procedure medications or intravascular contrast that cannot be adequately controlled with pre-medication.
15. Concurrent enrollment in another device or drug trial that has not completed the primary endpoint or clinically interferes with the current study endpoints. For patient previously participating in a drug trial, allow a wash-off period of at least 5 half-lives of the investigational drug.
16. Patient with significant co-morbid condition(s) which, at the discretion of the PI, are deemed to prohibit study entry.
17. Patient works the night shift.
18. Patient has valvular stenosis with risk of cardiac event with significant and/or abrupt decline in systolic blood pressure.
19. Untreated secondary cause of hypertension.
20. Device therapy within the past five years for the treatment of hypertension.
21. Prior renal stent or angioplasty.
22. Life expectancy <1 year.
23. Patients with history of renal transplant or planned renal transplantation within the next year.
24. History of one or more episodes of severe orthostatic hypotension within the past year.
25. Patient has unstable cardiac or pulmonary disease (including pulmonary hypertension) requiring chronic oxygen support.
26. Uncontrolled or inadequately treated bleeding diathesis.
27. Evidence of active infection within 7 days of procedure

Angiographic Exclusion Criteria

The following characteristics identified either on the renal artery CT scan or on the Eligibility II Renal artery Angiogram will prevent the patient from being included:

1. Main renal arteries < 4 mm in lumen diameter or < 20 mm in length; accessory renal arteries, if present, < 4 mm in lumen diameter or <10 mm in length.
2. Aorto-renal angle that in the operator's opinion prevents a safe cannulation of the renal artery.
3. Severe common femoral artery, common and/or external iliac artery, renal, iliac or aortic calcification or tortuosity that may compromise the safe performance and completion of the TIVUS™ procedure.
4. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the operator's opinion, would interfere with safe cannulation of the renal artery or meets local standards for surgical repair or interventional dilation (NOTE: vessel areas with calcification and fibromuscular dysplasia (FMD) should be avoided as intended treatment areas).
5. Any renal artery stenosis > 30% by visual assessment.
6. Any renal artery aneurysm (>50% of the main renal artery reference vessel diameter by visual estimate).
7. Presence of fibromuscular dysplasia
8. Significant renal artery atheroma, aneurysm, calcification in the target vessel identified on CT Angiogram

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | from baseline to 1 month post procedure
  acute treatment related adverse events including including all-cause mortality, acute kidney injury, significant embolic event, renal artery perforation or dissection requiring intervention, vascular complications, stroke, myocardial infarction, or transient ischemic attack, deterioration in renal function end-stage renal failure, hospital admission for hypertensive crisis not related to confirmed nonadherence with medications or the protocol, new renal artery stenosis of more than 70% and major access site complications or cardiovascular complications
Incidence of Adverse Events | from baseline to 12 month post procedure
  chronic treatment related adverse events including including all-cause mortality, acute kidney injury, significant embolic event, renal artery perforation or dissection requiring intervention, vascular complications, stroke, myocardial infarction, or transient ischemic attack, deterioration in renal function end-stage renal failure, hospital admission for hypertensive crisis not related to confirmed nonadherence with medications or the protocol, new renal artery stenosis of more than 70% and major access site complications or cardiovascular complications
Change in mean daytime ambulatory systolic BP | From baseline to 3 months post procedure
  Reduction in daytime ambulatory mean systolic blood pressure from baseline to 3 months after the procedure.

SECONDARY OUTCOMES:
Change in mean 24-hr ambulatory systolic and diastolic bp | 3, 6, 12, 24, 36 months
  Reduction of 24-hour ambulatory mean systolic and diastolic blood pressure from baseline
Change in mean 24-hr ambulatory diastolic bp | 3 months
  Reduction of 24-hour ambulatory mean diastolic blood pressure from baseline
Change in mean daytime ambulatory systolic bp | 6, 12, 24, 36 months
  Reduction of daylight ambulatory mean systolic blood pressure from baseline
Change in mean nighttime ambulatory systolic and diastolic bp | 3, 6, 12, 24, 36 months
  Reduction of nighttime ambulatory mean systolic and diastolic blood pressure from baseline
Change in mean office systolic and diastolic BP | 3, 6, 12, 24, 36 months
  Reduction of office mean systolic and diastolic blood pressure from baseline
Change in mean 24-hr ambulatory pulse | 3, 6, 12, 24, 36 months
  Reduction in mean 24-hour ambulatory pulse pressure from baseline
Rate of patients achieving target 24-hr ambulatory mean systolic BP | 3, 6, 12, 24, 36 months
  Number of patients achieving target 24-hour ambulatory mean systolic blood pressure (<130 mm Hg)
Rate of patients achieving target office systolic BP | 3, 6, 12, 24, 36 months
  Number of patients achieving target office systolic blood pressure (<140 mm Hg)
Change in number of antihypertensive medications taken | 6, 12 months
  Reduction in the number of antihypertensive medications taken and/or the dose taken
Percentage of patients who respond to treatment | 3, 6, 12 months
  Percentage of patients who respond to the treatment, with response defined as a reduction of at least 10mm in mean 24-hour ambulatory systolic blood pressure
Incidence of hypertensive or hypotensive emergency episodes | 3, 6, 12 months
  Incidence of hypertensive or hypotensive emergency episodes resulting in hospitalization
Change in renal function based on laboratory parameters | 3, 6, 12 months
  Changes in renal function, based on laboratory parameters such as eGFR (CKD-EPI) and serum creatinine
Change in renal function based on artery stenosis | 6, 12 months
  Changes in renal function, based on artery stenosis (>70%)
Incidence of heart failure | 3, 6, 12 months
  Episodes of heart failure events

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Principal Investigator — Columbia University/NYPH
Locations (9):
- United States (9):
  - Cardiology P.C., Birmingham, Alabama
  - ST Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Minneapolis Heart Institution Foundation, Minneapolis, Minnesota
  - Columbia University/NYPH, New York, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Medical University South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No